CLINICAL TRIAL: NCT01669668
Title: Radiofrequency Ablation Under Ideal Conditions in Hepatocellular Carcinoma
Brief Title: Radiofrequency Ablation in Treating Patients With Liver Cancer (Hepatocellular Carcinoma)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of referrals.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201207113
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA (Experimental): Patients undergo laparoscopic ultrasound followed by RFA.
  Interventions: Procedure: radiofrequency ablation; Procedure: laparoscopy

INTERVENTIONS:
Procedure: radiofrequency ablation — Undergo RFA
Procedure: laparoscopy — Undergo laparoscopic ultrasound

SUMMARY:
This phase II trial studies how effectively radiofrequency ablation prevents recurrence of hepatocellular carcinoma (HCC) in patients with easily removable tumors. Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HCC or unambiguous radiologic findings consistent with HCC (> 1 cm tumor with arterial hypervascularity and venous or delayed phase washout) in patients with underlying liver disease.
* Disease must be considered unresectable (as defined by protocol).
* Age between 18 and 69 (inclusive).
* Karnofsky performance status of ≥ 80%
* Normal organ and marrow function as defined below:
* leukocytes ≥3,000/mcL
* absolute neutrophil count ≥1,500/mcL
* platelets >100,000/mcL
* total bilirubin <2.0 mg/dL
* AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Presence of ≤ 3 tumors, all of which are ≤ 3 cm in size. This will be determined preoperatively and confirmed by intraoperative ultrasound.
* Liver function of Child-Pugh class A or B
* Tumor(s) must be more than 2 cm away from of major biliary duct or major blood vessel defined as the main portal vein and its right and left primary branches and the first 1 cm of the secondary branches of the common hepatic duct and its right and left primary branches or the first 1 cm of its secondary branches.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Hepatic tumor(s) with satellite lesions. A satellite lesion is defined as a tumor which is within 2 cm of the tumor being assessed for treatment and which has a diameter of less than 33% of the diameter of the tumor being assessed for treatment.
* Evidence of metastatic/extrahepatic disease based on abdominal and chest CT performed within 4 weeks of the procedure.
* Extrahepatic disease upon laparoscopy performed at the time of RFA. If extrahepatic disease is discovered at this laparoscopy, RFA will not be performed, and the patient will be considered ineligible for this study and will be replaced.
* Pregnancy. All women of childbearing potential must have a negative pregnancy test prior to enrollment in the study.
* Significant portal hypertension based on evidence of esophageal varices or ascites. Minimal portal hypertension or ascites will not be an exclusion criterion.
* Previous history of HCC or any other non-cutaneous malignancy.

Patients who are found to be ineligible due to intraoperative findings will be recorded as to the cause of ineligibility. They will not be counted as accrued patients.

-Inclusion of Women and Minorities Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Local recurrence, defined as the recurrence at the size of original tumor | Up to 2 years
  Local recurrence will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Morbidity and mortality associated with RFA under ideal conditions | 30 days
  The incidences of surgical complications and procedure-related death will be calculated.
Overall survival rate | At 2 years
  Kaplan-Meier product limit method will be used to estimate the 2-year overall survival. The median overall survival will also be
Disease-free survival rate | At 2 years
  Kaplan-Meier product limit method will be used to estimate the 2-year disease-free survival. The median disease-free survival will also be estimated.
Ability of patients who develop recurrence to undergo salvage transplantation | Up to 2 years
  At the time of recurrence, the patient is evaluated to see if she/he falls within the Milan criteria; if she/he does, then she/he is considered able to undergo salvage transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Strasberg, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu